CLINICAL TRIAL: NCT01785069
Title: A Prospective Multicenter Study of the Safety and Effectiveness of NATRELLE® 410 Highly Cohesive Anatomically Shaped Silicone-filled X-style and L-style Breast Implants
Brief Title: Safety and Effectiveness of NATRELLE® 410 Highly Cohesive, Anatomically Shaped, Silicone-filled X-Style and L-Style Breast Implants
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: There was no indication that long-term follow-up would differ between any of the studies that have evaluated devices within the 410 Style Matrix.
Sponsor: Allergan (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 410XL-001
Record Dates: First submitted 2013-01-14; First posted 2013-02-06 (Estimated); Results first posted 2020-06-25 (Actual); Last update posted 2020-06-25 (Actual); Status verified 2020-06

CONDITIONS: Breast Augmentation; Breast Reconstruction; Breast Implant Revision

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Device: Yes

ARMS (4):
- Augmentation (Experimental): Women who had breast augmentation with NATRELLE® 410 implants.
  Interventions: Device: Anatomically shaped, silicone-filled breast implants with low projection or extra-full projection
- Reconstruction (Experimental): Women who had breast reconstruction with NATRELLE® 410 implants.
  Interventions: Device: Anatomically shaped, silicone-filled breast implants with low projection or extra-full projection
- Revision-Augmentation (Experimental): Women who had revision of a previous breast augmentation with NATRELLE® 410 implants.
  Interventions: Device: Anatomically shaped, silicone-filled breast implants with low projection or extra-full projection
- Revision-Reconstruction (Experimental): Women who had revision of a previous breast reconstruction with NATRELLE® 410 implants.
  Interventions: Device: Anatomically shaped, silicone-filled breast implants with low projection or extra-full projection

INTERVENTIONS:
Device: Anatomically shaped, silicone-filled breast implants with low projection or extra-full projection — Surgical implant
  Other Names: NATRELLE® 410 Highly Cohesive, Anatomically Shaped, Silicone-Filled Breast Implants

SUMMARY:
This is a prospective, multicenter study of the safety and effectiveness of NATRELLE® 410 Highly Cohesive, Anatomically Shaped, Silicone-Filled X-Style and L-Style Breast Implants.

ELIGIBILITY:
Inclusion Criteria:

For entry in this study, participants must have been enrolled in the 410 Continued Access (CA) Clinical Study or 410 Continued Access Reconstruction/Revision Expansion (CARE) Clinical Study under the inclusion criteria listed below and received NATRELLE® 410 Highly Cohesive, Anatomically Shaped, Silicone-Filled X-Styles or L-Styles breast implants

* Female, age 18 or older
* Present with 1 or more of the following conditions:

  1. Primary breast augmentation (i.e., no previous breast implant surgery) indicated for subject dissatisfaction with size or shape of breast (e.g., mammary hypoplasia), asymmetry, ptosis, or aplasia
  2. Primary breast reconstruction (i.e., no previous breast implant surgery other than implantation of tissue expanders or contralateral augmentation for asymmetry) indicated, in the affected breast, for mastectomy for cancer, prophylactic mastectomy, or breast trauma (resulting in mastectomy) and for the unaffected breast, contralateral asymmetry (may be performed on the date of the mastectomy or the date when the permanent implants are placed in the reconstructed breast)
  3. Breast implant revision surgery (i.e., removal and replacement of breast implants) indicated for previous augmentation or reconstruction with silicone-filled or saline-filled breast implants
* Has adequate tissue available to cover implants
* Willing to undergo magnetic resonance imaging (MRI) at the specified follow-up visits for subjects at MRI designated sites and be eligible for MRI (e.g., no implanted metal or metal devices, no history of severe claustrophobia)

Exclusion Criteria:

For entry in this study, participants must have been enrolled in the 410 CA Clinical Study or 410 CARE Clinical Study, meeting the exclusion criteria listed below, did not receive any NATRELLE® 410 Highly Cohesive, Anatomically Shaped, Silicone-Filled FM, FF, MM, or MF Style Breast Implants, and have not undergone implant removal with or without replacement surgery

* Does not have advance fibrocystic disease considered to be premalignant without accompanying subcutaneous mastectomy
* Does not have existing carcinoma of the breast, without mastectomy
* Does not have abscess or infection in the body at the time of enrollment
* Is not pregnant or nursing
* Does not have any disease, including uncontrolled diabetes (e.g., hemoglobin A1c (HbA1c) > 8%), that is clinically known to impact wound healing ability
* Does not show tissue characteristics that are clinically incompatible with mammaplasty, such as tissue damage resulting from radiation inadequate tissue, compromised vascularity, or ulceration
* Does not have or is under treatment for any condition that may constitute an unwarranted surgical risk (e.g., unstable cardiac or pulmonary problems)
* Does not show psychological characteristics that may be incompatible with the surgical procedure and the prosthesis, such as inappropriate attitude or motivation (e.g., body dysmorphic disorder)
* Is not willing to undergo further surgery for revision, if medically required

Min Age: 18 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 355 (Actual)
Dates: Start 2012-12-10 (Actual); Primary Completion 2015-11-30 (Actual); Study Completion 2015-11-30 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Andrew Schumacher, Study Chair — Allergan
Locations (29):
- United States (29):
  - Laurence Berkowitz, Campbell, California
  - Roy Hong, Palo Alto, California
  - Eric Bachelor, Pleasanton, California
  - Gregory Liebscher, Colorado Springs, Colorado
  - Scott Spear, Washington D.C., District of Columbia
  - Calvin Peters, Orlando, Florida
  - Walter Erhardt, Albany, Georgia
  - James Namnoum, Atlanta, Georgia
  - Janet Turkle, Carmel, Indiana
  - Julene Samuels, Louisville, Kentucky
  - Timothy Mickel, Monroe, Louisiana
  - John Renucci, Grand Rapids, Michigan
  - Steven Morris, Midland, Michigan
  - Charles Nathan, Chesterfield, Missouri
  - Herluf Jr. Lund, Chesterfield, Missouri
  - Patricia McGuire, Creve Coeur, Missouri
  - Perry Johnson, Omaha, Nebraska
  - Peter Hyans, Berkeley Heights, New Jersey
  - Peter Hetzler, Little Silver, New Jersey
  - Caroline Glicksman, Sea Girt, New Jersey
  - Tracy Pfeifer, Great Neck, New York
  - Lloyd Gayle, New York, New York
  - Raymond Isakov, Cleveland, Ohio
  - Craig Colville, Toledo, Ohio
  - Frank Barone, Toledo, Ohio
  - Mary Gingrass, Nashville, Tennessee
  - Patrick Maxwell, Nashville, Tennessee
  - Jeffrey Friedman, Houston, Texas
  - Thomas Blanchard, Newport News, Virginia

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Augmentation | Revision-Augmentation | Reconstruction | Revision-Reconstruction
Started | 107 | 76 | 104 | 68
Completed | 95 | 64 | 91 | 54
Not Completed | 12 | 12 | 13 | 14
Not completed — Implanted with nonstudy device | 1 | 2 | 1 | 0
Not completed — Death | 0 | 0 | 2 | 0
Not completed — Subject choice | 2 | 2 | 0 | 1
Not completed — Lost to Follow-up | 1 | 2 | 4 | 1
Not completed — Reason not Specified | 1 | 2 | 1 | 4
Not completed — Not evaluable | 7 | 4 | 5 | 8

BASELINE CHARACTERISTICS:
Population: Evaluable population was defined as all screened participants who satisfied all eligibility criteria documented on the eligibility form, entered the study, and had a Year 3 office visit and magnetic resonance imaging (MRI) within the window.
Groups:
- Total: Total of all reporting groups
Arm/Group | Augmentation | Revision-Augmentation | Reconstruction | Revision-Reconstruction | Total
Number analyzed (Participants) | 100 | 72 | 99 | 60 | 331
Age, Continuous [Mean (Full Range); unit: years] | 35.1 [19.0 to 60.0] | 48.3 [26.0 to 68.0] | 51.8 [28.0 to 69.0] | 54.7 [25.0 to 71.0] | 46.5 [19.0 to 71.0]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 100 | 72 | 99 | 60 | 331
  Male | 0 | 0 | 0 | 0 | 0

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Participants According to Investigator Satisfaction With Implants
Description: The investigator rated their satisfaction with the participant's breast implant for each breast on a 5-point scale (1=Definitely dissatisfied, 2=Somewhat dissatisfied,3=Neither satisfied or dissatisfied, 4=Somewhat satisfied, 5=Definitely satisfied). If there was a different response for the left and right breasts the worst response was used. The percentage of participants where the investigator responded: "Definitely satisfied" or "Somewhat satisfied" is reported.
Time Frame: 3 years (followup after implantation that occurred between 07 July 2009 and 01 January 2012)
Population: Participants from the Evaluable population, all screened participants who satisfied all eligibility criteria documented on the eligibility form, entered the study, and had a Year 3 office visit and MRI within the window, with data available for analysis.
Measure: Number; unit: percentage of participants
Arm/Group | Augmentation | Revision-Augmentation | Reconstruction | Revision-Reconstruction
Number analyzed (Participants) | 100 | 66 | 95 | 49
percentage of participants | 99.0 | 97.0 | 100.0 | 95.9

2. Primary Outcome: Percentage of Participants According to Participant Satisfaction With Implants
Description: The participant rated their satisfaction with the breast implant for each breast on a 5-point scale (1=Definitely dissatisfied, 2=Somewhat dissatisfied, 3=Neither satisfied or dissatisfied, 4=Somewhat satisfied, 5=Definitely satisfied). If there was a different response for the left and right breasts the worst response was used. The percentage of participants who responded: "Definitely satisfied" or "Somewhat satisfied" is reported.
Time Frame: 3 years (followup after implantation that occurred between 07 July 2009 and 01 January 2012)
Population: as for outcome 1
Measure: Number; unit: percentage of participants
Arm/Group | Augmentation | Revision-Augmentation | Reconstruction | Revision-Reconstruction
Number analyzed (Participants) | 99 | 66 | 95 | 49
percentage of participants | 99.0 | 95.5 | 94.9 | 91.8

3. Secondary Outcome: Percentage of Participants With Local Complications
Description: Kaplan-Meier risk rates (estimation of the percentage of participants) of developing local complications is presented. Local complications collected in the study were: Asymmetry, Breast Pain, Capsular contracture, Delayed wound healing, Fluid accumulation/seroma, Implant malposition, Implant palpability/visibility. Implant rupture, Infection, Ptosis, Redness, Swelling, Wrinkling/rippling and Other complications (calcifications on mammogram, thing of mastectomy flap, deformity and nipple stretching).
Time Frame: 5 years (followup after implantation that occurred between 07 July 2009 and 01 January 2012)
Population: Evaluable population was defined as all screened participants who satisfied all eligibility criteria documented on the eligibility form, entered the study, and had a Year 3 office visit and MRI within the window.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Augmentation | Revision-Augmentation | Reconstruction | Revision-Reconstruction
Number analyzed (Participants) | 100 | 72 | 99 | 60
percentage of participants
  Any complication | 9.05 [4.81 to 16.66] | 15.71 [9.03 to 26.58] | 15.28 [9.34 to 24.43] | 3.77 [0.95 to 14.33]
  Asymmetry | 1.00 [0.14 to 6.89] | 0.00 [0.00 to 0.00] | 3.03 [0.99 to 9.10] | 0.00 [0.00 to 0.00]
  Breast pain | 2.00 [0.50 to 7.76] | 0.00 [0.00 to 0.00] | 1.01 [0.14 to 6.95] | 2.00 [0.28 to 13.36]
  Capsular contracture | 3.05 [0.99 to 9.17] | 3.12 [0.78 to 12.01] | 4.40 [1.67 to 11.34] | 3.67 [0.93 to 13.99]
  Delayed wound healing | 0.00 [0.00 to 0.00] | 1.39 [0.20 to 9.45] | 0.00 [0.00 to 0.00] | 0.00 [0.00 to 0.00]
  Fluid accumulation/seroma | 0.00 [0.00 to 0.00] | 1.39 [0.20 to 9.45] | 0.00 [0.00 to 0.00] | 0.00 [0.00 to 0.00]
  Implant malposition | 3.00 [0.98 to 9.01] | 4.17 [1.36 to 12.36] | 4.04 [1.54 to 10.41] | 1.67 [0.24 to 11.25]
  Implant palpability/visibility | 0.00 [0.00 to 0.00] | 1.39 [0.20 to 9.45] | 0.00 [0.00 to 0.00] | 0.00 [0.00 to 0.00]
  Implant rupture | 3.09 [1.01 to 9.29] | 12.64 [5.12 to 29.38] | 2.16 [0.55 to 8.38] | 5.91 [1.91 to 16.94]
  Infection | 0.00 [0.00 to 0.00] | 1.39 [0.20 to 9.45] | 2.02 [0.51 to 7.84] | 0.00 [0.00 to 0.00]
  Ptosis | 0.00 [0.00 to 0.00] | 1.39 [0.20 to 9.45] | 0.00 [0.00 to 0.00] | 0.00 [0.00 to 0.00]
  Redness | 1.00 [0.14 to 6.89] | 0.00 [0.00 to 0.00] | 2.02 [0.51 to 7.84] | 0.00 [0.00 to 0.00]
  Swelling | 1.05 [0.15 to 7.24] | 0.00 [0.00 to 0.00] | 0.00 [0.00 to 0.00] | 0.00 [0.00 to 0.00]
  Wrinkling/rippling | 0.00 [0.00 to 0.00] | 2.78 [0.70 to 10.65] | 0.00 [0.00 to 0.00] | 1.67 [0.24 to 11.25]
  Other complications | 1.00 [0.14 to 6.89] | 2.78 [0.70 to 10.65] | 2.12 [0.53 to 8.22] | 0.00 [0.00 to 0.00]

4. Secondary Outcome: Percentage of Participants With Reoperations
Description: Kaplan-Meier risk rates (estimation of the percentage of participants) of reoperation is reported.
Time Frame: 5 years (followup after implantation that occurred between 07 July 2009 and 01 January 2012)
Population: as for outcome 3
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Augmentation | Revision-Augmentation | Reconstruction | Revision-Reconstruction
Number analyzed (Participants) | 100 | 72 | 99 | 60
percentage of participants | 9.07 [4.82 to 16.71] | 25.64 [16.44 to 38.66] | 39.84 [30.88 to 50.30] | 39.01 [27.81 to 52.78]

5. Secondary Outcome: Percentage of Participants With Implant Removal With or Without Replacement
Description: Kaplan-Meier risk rates (estimation of the percentage of participants) of implant removal with or without replacement
Time Frame: 5 years (followup after implantation that occurred between 07 July 2009 and 01 January 2012)
Population: as for outcome 3
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Augmentation | Revision-Augmentation | Reconstruction | Revision-Reconstruction
Number analyzed (Participants) | 100 | 72 | 99 | 60
percentage of participants | 1.05 [0.15 to 7.24] | 12.42 [4.43 to 32.13] | 2.35 [0.59 to 9.08] | 6.13 [1.98 to 18.16]

ADVERSE EVENTS:
Time Frame: 5 years (followup after implantation that occurred between 07 July 2009 and 01 January 2012)
Description: Adverse events were not collected in this study. Deaths are reported as Serious Adverse Events. Specific local complications were collected and are reported in the Outcome Measure section. Evaluable population.
Arm/Group | Augmentation | Reconstruction | Revision-Augmentation | Revision-Reconstruction
Serious Adverse Events (participants affected / at risk) | 0/100 | 2/72 | 0/99 | 0/60
Other Adverse Events (participants affected / at risk) | 0/0 | 0/0 | 0/0 | 0/0
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Augmentation (N=100) | Reconstruction (N=72) | Revision-Augmentation (N=99) | Revision-Reconstruction (N=60)
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0 | 0 — Following knee surgery
Bacterial pneumonia (Infections and infestations) | 0 | 1 | 0 | 0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
A disclosure restriction on the PI is that the sponsor can review results communications prior to public release and can embargo communications regarding trial results for a period that is less than or equal to 90 days from the time submitted to the sponsor for review. The sponsor cannot require changes to the communication and cannot extend the embargo.